CLINICAL TRIAL: NCT00126945
Title: A Primary Vaccination Study to Assess the Immunogenicity, Safety & Reactogenicity of 1 Dose of 4 Different Formulations of GSK Biologicals' Meningococcal Conjugate Vaccine (MenACWY) vs 1 Dose of MENCEVAX™ ACWY in Healthy Subjects Aged 15-19 Years
Brief Title: Evaluate 4 Different Formulations of Meningococcal Serogroups A,C,W-135,Y Conjugate Vaccine When Given as 1 Dose to Healthy Subjects Aged 15-19 Yrs
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 104702
Record Dates: First submitted 2005-08-04; First posted 2005-08-05 (Estimated); Last update posted 2016-09-21 (Estimated); Status verified 2016-09

CONDITIONS: Infections, Meningococcal
Keywords: Meningococcal serogroups A, C, W-135, Y disease
MeSH Terms: conditions — Meningococcal Infections | interventions — Meningococcal Vaccines

INTERVENTIONS:
Biological: Meningococcal Vaccine

SUMMARY:
The purpose of this study is to evaluate the immunogenicity, safety and reactogenicity of one dose of four different formulations of the MenACWY conjugate vaccine when given to healthy subjects aged 15-19 years. The selection of the best formulation will be based on data obtained up to one month after the vaccine dose.

DETAILED DESCRIPTION:
The study is open. However, the 4 different formulations of GSK's MenACWY conjugate vaccine will be administered in a double-blind manner. Mencevax™ ACWY vaccine will serve as active control. Subjects will receive one vaccine dose only (GSK's MenACWY conjugate vaccine or Mencevax™ ACWY vaccine), and will have 2 blood samples taken, before and one month after vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female between, and including, 15 and 19 years of age at the time of vaccination.
* Subject with previously completed routine childhood vaccinations to the best of his/her knowledge or his/her parents'/guardians' knowledge.
* Female subjects should be of non-childbearing potential.

Exclusion Criteria:

* Previous vaccination against OR history of OR exposure within previous 12 months to meningococcal serogroup A, C, W-135 or Y disease.
* Administration of a tetanus vaccine within 6 months before study vaccination.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus (HIV) infection.
* A family history of congenital or hereditary immunodeficiency.
* History of any neurologic disorders or seizures.

Ages: 15 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 125 (Actual)
Dates: Start 2005-08; Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
Percentage of serum bactericidal activity SBA-MenA, SBA-MenC, SBA-MenW-135 and SBA-MenY responders (i.e. 4-fold increase in serum bactericidal antibody [SBA] titre from pre to post vaccination) at 1 month after the first vaccine dose

SECONDARY OUTCOMES:
Antibodies to MenACWY before + 1 m after dose 1, 12 m after dose 1 in control + with selected vaccine groups, 1 m after booster
Solicited, unsolicited symptoms after each dose and serious adverse events (SAEs)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Aarhus N, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Ostergaard L, Lebacq E, Poolman J, Maechler G, Boutriau D. Immunogenicity, reactogenicity and persistence of meningococcal A, C, W-135 and Y-tetanus toxoid candidate conjugate (MenACWY-TT) vaccine formulations in adolescents aged 15-25 years. Vaccine. 2009 Jan 1;27(1):161-8. doi: 10.1016/j.vaccine.2008.08.075. Epub 2008 Oct 1. PMID 18834910
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 104702 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 104702 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 104702 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 104702 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 104702 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 104702 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register